CLINICAL TRIAL: NCT05308121
Title: Investigation of Trimester-Specific Normative Values of Biomechanical and Viscoelastic Properties of Achilles Tendon in Pregnant Women-Pilot Study
Brief Title: Biomechanical and Viscoelastic Properties of Achilles Tendon in Pregnant Women-Pilot Study
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 20
Record Dates: First submitted 2022-03-12; First posted 2022-04-01 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pregnant Women
Keywords: pregnant women; achilles tendon; stiffness; creep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First trimester pregnant women (first pregnancy): This group will consist of women in the first trimester of pregnancy. Pregnant women will be evaluated 2 points of the Achilles Tendon
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Achilles tendon; Other: Evaluation of foot characteristics
- Second trimester pregnant women (first pregnancy): This group will consist of women in the second trimester of pregnancy. Pregnant women will be evaluated 2 points of the Achilles Tendon
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Achilles tendon; Other: Evaluation of foot characteristics
- Third trimester pregnant women (first pregnancy): This group will consist of women in the third trimester of pregnancy. Pregnant women will be evaluated 2 points of the Achilles Tendon
  Interventions: Other: Evaluation of biomechanics and viscoelastic properties of Achilles tendon; Other: Evaluation of foot characteristics

INTERVENTIONS:
Other: Evaluation of biomechanics and viscoelastic properties of Achilles tendon — The biomechanical and viscoelastic properties of the Achilles tendon will be measured in the side lying position. Measurements will be taken from two different points with the ankle in the neutral position.
Other: Evaluation of foot characteristics — The mobility of foot, morphological changes of foot and foot posture will be evaluated

SUMMARY:
There is anatomical fascial continuity and functional connection between the plantar fascia, which has important roles in foot biomechanics, and the fibers of the Achilles tendon, and the change that will occur in any of these tissues is reflected in the other. However, it has not been objectively clarified how the tissue properties of the Achilles tendon, which plays an important role in foot biomechanics, such as the plantar fascia, change with pregnancy. Therefore, the aim of this pilot study is to investigate the trimester-specific biomechanical (stiffness, decrement and tone) and viscoelastic (creep and relaxation time) properties of the Achilles tendon, which adapts to changes in the foot structure during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* First pregnancy
* They are between the ages of 18-40
* Pre-pregnancy Body-Mass-Index (BMI) < 30 kg/m2

Exclusion Criteria:

* Presence of any connective tissue disease that would affect the biomechanical or viscoelastic properties of the fascia
* Deterioration of skin integrity in measurement areas
* Presence of orthopedic, neurological, rheumatic problems that may cause musculoskeletal disorders and deviations from normal in biomechanical alignment
* History of surgery or fracture in the lower extremity and foot-ankle region in the last 6 months
* Defining metabolic disorders such as type I, II diabetes, gestational diabetes mellitus (GDM), preeclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women (first pregnancy)
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of biomechanical properties of achilles tendon | Measurement the baseline stiffness values of Achilles tendon between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the stiffness (N/m) of the achilles tendon (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of biomechanical properties of achilles tendon | Measurement the baseline decrement values of Achilles tendon between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the decrement of the achilles tendon (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of biomechanical properties of achilles tendon | Measurement the baseline tone values of Achilles tendon between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the tone (Hz) of the achilles tendon (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of viscoelastic properties of achilles tendon | Measurement the baseline creep values of Achilles tendon between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the creep of the achilles tendon (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.
Evaluation of viscoelastic properties of achilles tendon | Measurement the baseline relaxation time values of Achilles tendon between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the relaxation time (ms) of the achilles tendon (with MyotonPro, Myoton AS, Tallin, Estonia) in the side lying position.

SECONDARY OUTCOMES:
Evaluation of Body Weight | Measurement the baseline body weight (kg) between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Measuring of the Body Weight
Evaluation of Body Mass Index (BMI) | Measurement the baseline BMI values at between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  BMI (kg/m2) will be calculated as person's weight in kilograms divided by the square of height in meters.
Evaluation of foot mobility | The measurement of the baseline navicular drop values between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Navicular drop values will be measured
Evaluation of foot morphological properties | The measurement of the baseline foot length between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Foot length will be measured
Evaluation of foot morphological properties | The measurement of the baseline foot width between 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Foot width will be measured
Evaluation of foot posture | The measurement of the baseline foot posturebetween 10-14 weeks, between 20-24 weeks and between 32-36 weeks.
  Foot posture will be evaluated according to foot posture index

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dumas GA, Reid JG. Laxity of knee cruciate ligaments during pregnancy. J Orthop Sports Phys Ther. 1997 Jul;26(1):2-6. doi: 10.2519/jospt.1997.26.1.2. PMID 9201635
- [Result] Marnach ML, Ramin KD, Ramsey PS, Song SW, Stensland JJ, An KN. Characterization of the relationship between joint laxity and maternal hormones in pregnancy. Obstet Gynecol. 2003 Feb;101(2):331-5. doi: 10.1016/s0029-7844(02)02447-x. PMID 12576258
- [Result] Orner S, Kratzer W, Schmidberger J, Gruner B. Quantitative tissue parameters of Achilles tendon and plantar fascia in healthy subjects using a handheld myotonometer. J Bodyw Mov Ther. 2018 Jan;22(1):105-111. doi: 10.1016/j.jbmt.2017.06.015. Epub 2017 Jun 21. PMID 29332731
- [Result] Snow SW, Bohne WH, DiCarlo E, Chang VK. Anatomy of the Achilles tendon and plantar fascia in relation to the calcaneus in various age groups. Foot Ankle Int. 1995 Jul;16(7):418-21. doi: 10.1177/107110079501600707. PMID 7550955
- [Result] Chang TT, Feng YN, Zhu Y, Liu CL, Wang XQ, Zhang ZJ. Objective Assessment of Regional Stiffness in Achilles Tendon in Different Ankle Joint Positions Using the MyotonPRO. Med Sci Monit. 2020 Oct 19;26:e926407. doi: 10.12659/MSM.926407. PMID 33071278